CLINICAL TRIAL: NCT02738697
Title: The Clinical Randomized Trial of Adjuvant Chemotherapy With FOLFOX in HCC Patients at High Risk After Resection
Brief Title: Adjuvant Chemotherapy With FOLFOX in HCC Patients After Resection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rong-ping Guo, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSUCC-HCC-ADCHEMO
Record Dates: First submitted 2016-03-24; First posted 2016-04-14 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Carcinoma, Hepatocellular
Keywords: Carcinoma,Hepatocellular; Adjuvant chemotherapy; Microvessels invasion; Survival; Recurrence
MeSH Terms: conditions — Carcinoma, Hepatocellular; Recurrence | interventions — Chemotherapy, Adjuvant; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adjuvant chemotherapy (Experimental): 8~12 cycles of adjuvant chemotherapy with FOLFOX were performed 4-6 weeks after radical surgery
  Interventions: Drug: Adjuvant chemotherapy
- Follow-up (Other): Routine follow-up were performed instead of adjuvant chemotherapy
  Interventions: Procedure: Follow-up

INTERVENTIONS:
Drug: Adjuvant chemotherapy — 8~12 cycles of adjuvant chemotherapy with FOLFOX were performed 4-6 weeks after radical surgery
  Other Names: adjuvant chemotherapy with FOLFOX
  Arms: Adjuvant chemotherapy
Procedure: Follow-up — Patients received just follow-up instead of adjuvant chemotherapy
  Arms: Follow-up

SUMMARY:
Hepatocellular carcinoma (HCC) is the sixth most common malignancies worldwide and the second leading cause of cancer-related death. Surgical resection is still the main radical approach for HCC, but the recurrence rate after hepatectomy is very high, which hampers the further improvement of prognosis of HCC patients. The conventional risk factors of recurrence including: huge tumor, multiple lesions, vessels invasion and tumor rupture. Recently, the microvessels invasion (MVI) has been recognized a novel risk factor of recurrence after hepatectomy. The investigators' previous study showed that the recurrence rate is more than 50% for the patients with >5cm solitary tumor and MVI. The MVI was confirmed as the only independent risk factor for the overall and disease-free survival of HCC patients in multiple variables analysis. It is important to reduce the recurrence and prolong the survival of patients after hepatectomy with effective adjuvant therapy. Reported at 2014 American Society of Clinical Oncology (ASCO) annual meeting, A phase III randomized, double-blind, placebo-controlled trial of adjuvant sorafenib after resection or ablation to prevent recurrence of hepatocellular carcinoma (STORM trial) failed to meet the primary endpoint-recurrence free survival (RFS). Given the inspiring result of a recent trial, which compared with single agent of doxorubicin, the oxaliplatin-containing regimens (FOLFOX) showed significant improvement in OS, objective response rate (ORR) and disease control rate (DCR) in Asian (especially China) HCC patients. Based on these rationales, the investigators design the current prospective randomized clinical trial to evaluate the effect of adjuvant chemotherapy with FOLFOX to prolong the overall survival and reduce the recurrence in HCC patients at high risk (>5cm solitary tumor and MVI) after resection, compared to vigilant follow-up.

DETAILED DESCRIPTION:
The patients with solitary tumor more than 5cm and microvessels invasion after radical hepatectomy were randomized to receive adjuvant FOLFOX chemotherapy （8~12 cycles) or follow-up. The main endpoint: overall survival (OS), disease-free survival(DFS) and safety were compared between this two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18~75 years;
2. Eastern Cooperative Oncology Group performance status (ECOG PS) score <=2;
3. Histologically confirmed hepatocellular carcinoma with microvessels invasion;
4. No previous treatment for HCC;
5. More than 5 cm solitary tumor before surgery confirmed by more than 2 radiological examinations;
6. R0 resection achieved;
7. No recurrence evidence in radiological follow-up 3~5 weeks after surgery;
8. Adequate hematologic parameters and liver and kidney functions: (1) Neutrophils Absolute >=1.5*10^9/L; (2) Hemoglobin >=90g/L; (3) Platelet count >=75*10^9/L; (4) Serum albumin >=35g/L; (5) Serum total bilirubin <=1.5*upper limit of normal (ULN); (6) Serum Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) <2.5*ULN; (7) Serum creatinine <=1.5*ULN; (8) International normalized ratio (INR)<=1.5;
9. Give signed informed consent before enrollment.

Exclusion Criteria:

1. Function impairment of vital organs (heart, lung, kidney, etc), serious infection or >grade 2 adverse events (Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0);
2. Histologically confirmed of positive resection margin (R1 resection);
3. Previous or current malignant tumor beyond HCC;
4. Allergy to any agent of the FOLFOX regimen;
5. History of organ transplantation;
6. Previously receiving other treatments for HCC;
7. Pregnant or breastfeeding women, and women of childbearing potential without adequate contraception;
8. Neurological or mental abnormalities that may affect cognitive assessment and inform consent;
9. Concomitant anti-tumor therapy or participating in other interventional clinical trials;
10. Other psychological, family or social reason, which would affect compliance with the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  The overall survival is defined as the percentage of patients who are alive at 5 years after their enrollments of this study.

SECONDARY OUTCOMES:
Disease-free survival | 5 years
  The disease-free survival is defined as the percentage of patients who are alive at 5 years without any signs or symptoms of HCC after their enrollments of this study.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | 5 years
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Rong-Ping Guo, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- SUN YAT-SEN University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qin S, Cheng Y, Liang J, Shen L, Bai Y, Li J, Fan J, Liang L, Zhang Y, Wu G, Rau KM, Yang TS, Jian Z, Liang H, Sun Y. Efficacy and safety of the FOLFOX4 regimen versus doxorubicin in Chinese patients with advanced hepatocellular carcinoma: a subgroup analysis of the EACH study. Oncologist. 2014 Nov;19(11):1169-78. doi: 10.1634/theoncologist.2014-0190. Epub 2014 Sep 15. PMID 25223462
- [Result] Qin S, Bai Y, Lim HY, Thongprasert S, Chao Y, Fan J, Yang TS, Bhudhisawasdi V, Kang WK, Zhou Y, Lee JH, Sun Y. Randomized, multicenter, open-label study of oxaliplatin plus fluorouracil/leucovorin versus doxorubicin as palliative chemotherapy in patients with advanced hepatocellular carcinoma from Asia. J Clin Oncol. 2013 Oct 1;31(28):3501-8. doi: 10.1200/JCO.2012.44.5643. Epub 2013 Aug 26. PMID 23980077
- [Result] Llovet JM, Ricci S, Mazzaferro V, Hilgard P, Gane E, Blanc JF, de Oliveira AC, Santoro A, Raoul JL, Forner A, Schwartz M, Porta C, Zeuzem S, Bolondi L, Greten TF, Galle PR, Seitz JF, Borbath I, Haussinger D, Giannaris T, Shan M, Moscovici M, Voliotis D, Bruix J; SHARP Investigators Study Group. Sorafenib in advanced hepatocellular carcinoma. N Engl J Med. 2008 Jul 24;359(4):378-90. doi: 10.1056/NEJMoa0708857. PMID 18650514
- [Result] Llovet JM, Di Bisceglie AM, Bruix J, Kramer BS, Lencioni R, Zhu AX, Sherman M, Schwartz M, Lotze M, Talwalkar J, Gores GJ; Panel of Experts in HCC-Design Clinical Trials. Design and endpoints of clinical trials in hepatocellular carcinoma. J Natl Cancer Inst. 2008 May 21;100(10):698-711. doi: 10.1093/jnci/djn134. Epub 2008 May 13. PMID 18477802
- [Result] Bruix J, Takayama T, Mazzaferro V, Chau GY, Yang J, Kudo M, Cai J, Poon RT, Han KH, Tak WY, Lee HC, Song T, Roayaie S, Bolondi L, Lee KS, Makuuchi M, Souza F, Berre MA, Meinhardt G, Llovet JM; STORM investigators. Adjuvant sorafenib for hepatocellular carcinoma after resection or ablation (STORM): a phase 3, randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2015 Oct;16(13):1344-54. doi: 10.1016/S1470-2045(15)00198-9. Epub 2015 Sep 8. PMID 26361969